CLINICAL TRIAL: NCT05368207
Title: Pembrolizumab in Small Cell Carcinoma of Ovary - Hypercalcemic Type Patient (Pemb-HT)
Brief Title: Pembrolizumab in Small Cell Carcinoma of Ovary - Hypercalcemic Type Patient
Acronym: Pemb-HT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pemb-HT
Record Dates: First submitted 2021-12-10; First posted 2022-05-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Small Cell Carcinoma, Hypercalcaemic Type; Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Small Cell; Ovarian Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: It is an open-label single patient Clinical Trial to be conducted at Princess Margaret Cancer Centre for a patient with Small Cell Carcinoma of Ovary - Hypercalcemic Type (SCCOHT) who has rare and aggressive malignancy with no current consensus on treatment approach and surveillance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be given as an intravenous infusion at 200 mg, every 6 weeks, for 6 cycles.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is an antineoplastic agent, monoclonal antibody against PD-L1.
  Other Names: KEYTRUDA

SUMMARY:
This is a study of pembrolizumab as consolidation therapy for a patient with small cell carcinoma of the ovary, hypercalcemic type (SCCOHT).

DETAILED DESCRIPTION:
It is an open-label single patient Clinical Trial to be conducted at Princess Margaret Cancer Centre for a patient with Small Cell Carcinoma of Ovary - Hypercalcemic Type (SCCOHT) who has rare and aggressive malignancy with no current consensus on treatment approach and surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with small cell carcinoma of the ovary, hypercalcemic type (SCCOHT)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Determined by CT scans

SECONDARY OUTCOMES:
overall performance status | 2 years
  Eastern cooperative oncology group (ECOG) score, patient-reported symptoms as well as objective measurements by CT scans.
Objective evidence of response to treatment | 2 years
  Recorded with CA-125 every 6 weeks and CT scans after every 2 cycles of treatment
Exploratory Endpoint | 2 Years
  Exploratory Endpoint will be measured by circulating DNA to monitor minimal residual disease

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No